CLINICAL TRIAL: NCT06670222
Title: Phase I Study With Dose-escalation and Expansion Evaluating the Safety and Efficacy of Oral Arsenic (ATO) in Low-risk Myelodysplastic Syndromes Failing Erythropoiesis Stimulating Agents and Luspatercept (or Ineligible for the Latter)
Brief Title: Oral Arsenic (ATO) in Low-risk Myelodysplastic Syndromes (MDS)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Groupe Francophone des Myelodysplasies (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATOMYELO; 2024-515311-22-00 (EU CTIS Number)
Record Dates: First submitted 2024-10-15; First posted 2024-11-01 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Low-risk Myelodysplastic Syndromes
Keywords: Oral Arsenic; Low-risk myelodysplastic syndromes
MeSH Terms: interventions — Arsenic Trioxide

STUDY DESIGN:
Intervention Model Description: Dose escalation cohort to determine the dose limiting toxicity according to a BOIN (Bayesian optimal interval) scheme. Three doses of oral Arsenic will be tested, and 9 patients will be treated at each dose.
  An expansion cohort at the selected dose will be conducted with 6 patients, for a maximum of 15 patients included at this dose level.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ATO (Experimental): Oral Arsenic treatment
  Interventions: Drug: Arsenic Trioxide (ATO)

INTERVENTIONS:
Drug: Arsenic Trioxide (ATO) — Study treatment: oral Arsenic 5d/7 for 21 days over a 28-day cycle, three doses tested (0.10 mg/kg, 0.15 mg/kg and 0.20 mg/kg).
  Dose escalation cohort to determine the dose limiting toxicity according to a BOIN (Bayesian optimal interval) scheme, 9 patients will be treated at each dose.
  An expansion cohort at the selected dose will be conducted with 6 patients.
  Tolerability will be assessed after one treatment cycle. Response will be assessed after 3 cycles of treatment. Responders may continue study treatment until progression or limiting toxicity. Limiting toxicity is defined as any grade III/IV extra-hematological toxicity or grade IV hematological toxicity lasting more than 25 days.

SUMMARY:
Phase I study with dose-escalation and expansion evaluating the safety and efficacy of oral Arsenic (ATO) in low-risk Myelodysplastic Syndromes having failed to Erythropoiesis Stimulating Agents and Luspatercept (or ineligible for the latter).

DETAILED DESCRIPTION:
Dose escalation cohort to determine the dose limiting toxicity according to a BOIN (Bayesian optimal interval) scheme.

Patients will receive one dose of study treatment (oral Arsenic (ATO)) 5d/7 for 21 days over a 28-day cycle.

Three doses of ATO will be tested (0.10 mg/kg, 0.15 mg/kg and 0.20 mg/kg), and 9 patients will be treated at each dose.

An expansion cohort at the selected dose based on DSMB recommendations will be conducted with 6 patients, for a maximum of 15 patients included at this dose level.

Tolerability will be assessed after one treatment cycle. Response will be assessed after 3 cycles of treatment. Responders may continue study treatment until progression or limiting toxicity. Limiting toxicity is defined as any grade III/IV extra-hematological toxicity or grade IV hematological toxicity lasting more than 25 days.

If there is no response, patients will stop treatment and enter the follow-up phase of the study.

ELIGIBILITY:
Inclusion criteria:

Patients must meet all the following criteria to participate in the study:

1. Myelodysplastic syndrome according to WHO (World Health Organization) 2022 classification
2. Age ≥ 18 years
3. Patient with low-risk Myelodysplastic Syndromes according to Revised International Prognostic Scoring System (IPSS-R) classification (very low, low, intermediate):

   * non-sideroblastic who failed to achieved a response or who subsequently relapse after Erythropoiesis Stimulating Agents (ESA) (at Epoetin alfa 60000UI or equivalent over at least 12 weeks) without disease progression or ineligible to ESA (defined by Erythopoietine (EPO) > 500UI/L)
   * sideroblastic who failed to achieved a response or who subsequently relapse after ESA (at Epoetin alfa 60000UI or equivalent over at least 12 weeks) or ineligible for ESA (defined by EPO >500UI/L) and who failed to achieved a response or who subsequently relapse after Luspatercept
   * del (5q) who failed to achieved a response or who subsequently relapse after ESA (at Epoetin alfa 60000IU or equivalent over at least 12 weeks) and who failed to achieved a response or who subsequently relapse after Lenalidomide
4. Transfusion dependence (at least 3 RBC (Red Blood Cell) within a 16-week period and at least 2 transfusion episodes during this period)
5. Patient not eligible for another clinical trial
6. Adequate renal function defined by creatinine level less than 1.5 times the upper limit of normal and creatinine clearance ≥ 40mL/min (according to MDRD (Modification of Diet in Renal Disease) formula)
7. Adequate liver function defined by total bilirubin and transaminases less than 1.5 times the upper limit of normal
8. Patient not refractory to platelet transfusions
9. Written consent
10. Patient must understand and voluntarily sign informed consent form
11. Patient must be able to adhere to the visit schedule as outlined in the study and follow protocol requirements
12. Performance status 0-2 at the time of screening
13. A FCBP (female of childbearing potential) for this study was defined as a sexually mature woman who: (1) had not undergone a hysterectomy or bilateral oophorectomy; or (2) had not been naturally postmenopausal (amenorrhea following cancer therapy did not rule out childbearing potential) for at least 24 consecutive months (ie, has had menses at any time in the preceding 24 consecutive months).

    A FCBP participating in the study must:
    * Have had 2 negative pregnancy tests as verified by the investigator prior to starting IP (unless the screening pregnancy test was done within 72 hours of Cycle 1 Day 1). She must have had agreed to ongoing a monthly pregnancy testing during the course of the study and after end of treatment.
    * If sexually active, agreed to have used, and been able to comply with, highly effective contraception** without interruption, 5 weeks prior to starting treatment, during treatment (including dose interruptions), and for 24 weeks after discontinuation of treatment.

      * Highly effective contraception was defined in this protocol as the following (information also appeared in the Informed Consent Form): Hormonal contraception (eg, birth control pills, injection, implant, transdermal patch, vaginal ring), intrauterine device, tubal ligation (tying your tubes), or a partner with a vasectomy.
14. Male subjects must: Have agreed to use a condom, defined as a male latex condom or nonlatex condom NOT made out of natural (animal) membrane (eg, polyurethane), during sexual contact with a pregnant female or a FCBP while participating in the study, during dose interruptions, and for at least 24 weeks following treatment discontinuation, even if he had undergone a successful vasectomy.

Exclusion criteria:

Any patient meeting one of the following criteria cannot be included in the study:

1. Severe infection or any uncontrolled severe condition
2. Uncontrolled hypertension
3. Significant cardiac disease - NYHA (New York Heart Association) Class III or IV or having suffered a myocardial infarction in the last 6 months
4. QTcF (Fridericia's corrected QT interval) > 460ms
5. Use of investigational agents within 30 days or any anticancer therapy (including IMiD (Immunomodulatory treatments)) within 2 weeks before the study entry with the exception of hydroxyurea. The patient must have recovered at least a grade 1 from all acute toxicity from any previous therapy. However, patients may have received Lenalidomide, hypomethylating agent, or anti-lymphocytic serum (ALS) (but not within 4 weeks before the study entry and, for ALS, within 16 weeks before the study entry).
6. Use of EPO within 4 weeks before the study entry
7. Active cancer or cancer during the year prior to trial entry other than basal cell carcinoma, or carcinoma in situ of the cervix or breast
8. Patient already enrolled in another therapeutic trial of an investigational drug
9. Known Human Immunodeficiency Virus infection or active hepatitis B or C
10. Women who are or could become pregnant or who are currently breastfeeding
11. Any medical or psychiatric contraindication that would prevent the patient from understanding and signing the informed consent form
12. Patient eligible for allogeneic stem cell transplantation
13. No affiliation to a health insurance system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-07-22 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
To determine the dose-limiting toxicity (DLT) of oral Arsenic (ATO) | At the end of cycle 1 (each cycle is 28 days)
  Dose-limiting toxicity will be defined by the occurrence during the first treatment cycle of any of the following toxicities related to the trial drug (oral ATO):
  * Non-hematological toxicity of grade ≥ 3
  * Hematological toxicity of grade ≥ 4 corresponding to a decrease of 50% or more of absolute neutrophil count (ANC) or platelet count from baseline or lower limit (if baseline was above normal), without recovery at D42 of the first cycle.

SECONDARY OUTCOMES:
To determine safety profile | Through study completion, an average of 2 years
  Toxicities measured according to CTCAE (Common Terminology Criteria for Adverse Events)
Pharmacokinetics | At the end of cycle 1 (each cycle is 28 days)
  Measurement of the peak plasma concentration (Cmax) of oral ATO
Pharmacokinetics | At the end of cycle 1 (each cycle is 28 days)
  Measurement of area under the plasma concentration versus time curve (AUC) for oral ATO
Pharmacokinetics | At the end of cycle 1 (each cycle is 28 days)
  Measurement of the residual concentration (Cmin) of oral ATO
Efficacy | At the end of cycle 3 (each cycle is 28 days)
  Response rate (Complete Response + Partial Response + stable disease with hematological improvement according to IWG (International Working Group) 2018 criteria)
Response duration | Through study completion, an average of 2 years
  Response duration measured from date of objective response to date of relapse or progression (or date of last news in absence of event)
Progression-free survival | Through study completion, an average of 2 years
  Rate and time to transformation to high-risk myelodysplastic syndrome (MDS) or Acute Myeloid Leukemia (AML)
Overall survival | Through study completion, an average of 2 years
  Overall survival from date of inclusion to death or date of last news

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CHU de Nice - Hôpital l'Archet - Service d'hématologie clinique, Nice
  - Hôpital Saint Louis - Service Hématologie séniors, Paris
  - Institut Gustave Roussy - Service d'hématologie, Villejuif

IPD SHARING:
Plan to Share IPD: No